CLINICAL TRIAL: NCT01649154
Title: Clinical Trial on Harmonic Focus Shears Versus Ligasure Small Jaw and Clamp-and-tie Technique for Total Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regina Apostolorum (Other)
Responsible Party: Principal Investigator, Giulia Cosenza, Principal Investigator, Ospedale Regina Apostolorum
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 8580/DS/CE
Record Dates: First submitted 2012-06-24; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-06

CONDITIONS: Benign Thoroid Disease Requiring Total Thyroidectomy
MeSH Terms: interventions — Cytidine Diphosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ligasure Small-JAW (Active Comparator)
  Interventions: Procedure: Total Thyroidectomy with cut and tie technique vs Total Thyroidectomy with Ligasure Small-JAW vs Total Thyroidectomy with Harmonic Focus
- Harmonic Focus (Active Comparator)
  Interventions: Procedure: Total Thyroidectomy with cut and tie technique vs Total Thyroidectomy with Ligasure Small-JAW vs Total Thyroidectomy with Harmonic Focus
- Clamp-and-Tie technique (Active Comparator)
  Interventions: Procedure: Total Thyroidectomy with cut and tie technique vs Total Thyroidectomy with Ligasure Small-JAW vs Total Thyroidectomy with Harmonic Focus

INTERVENTIONS:
Procedure: Total Thyroidectomy with cut and tie technique vs Total Thyroidectomy with Ligasure Small-JAW vs Total Thyroidectomy with Harmonic Focus

SUMMARY:
The Harmonic Focus and Ligasure small-Jaw are the last device designed for thyroid surgery. The aim is to assess: 1. decrease of operative time (minutes); 2. decrease of post-operative blood loss (milliliters); 3. decrease of post-operative stay (days); decrease of post-operative complications (%, hypocalcemia, laringeal nerve demage), compared to traditional dissection in a prospective randomized trial of total thyroidectomy procedures, for benign disease.

DETAILED DESCRIPTION:
A single-blinded prospective randomized controlled trial was conducted at a tertiary referral center. A total of 120 patients who required a thyroidectomy for thyroid benign disease, will be randomized to either Harmonic Focus or Ligasure small-Jaw or clamp-and-tie technique during thyroidectomy. The operative time (minutes), morbidity rate (%), post-operative blood loss (milliliters), hospital stay (days), post-operative hypocalcemia (%), and cost of thyroidectomy (euros) were compared between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* thyroid benign disease

Exclusion Criteria:

* malignant disease
* thyroid malign disease requiring lymphadenectomy
* coagulatory disease

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Improvement of post-operative outcomes (morbidity, hospital stay, costs) with new generation devices for total thyroidectomy.

SECONDARY OUTCOMES:
Cost assessment of new generation devices in thyroid surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regina Apostolorum, Albano Laziale, Rome, Italy